CLINICAL TRIAL: NCT01264497
Title: A Double-blind, Randomized, Parallel, Placebo-controlled 12-week Evaluation of the Safety of Two Doses of TH9507 in Subjects With Stable, Type 2 Diabetes Mellitus
Brief Title: Safety Study of TH9507 in Subjects With Stable, Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theratechnologies (Industry)
Responsible Party: Bruno Lussier/Medical Director, Theratechnologies
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH9507/II/Diabetes/006
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TH9507 — 1 and 2 mg, sc daily for 12 weeks

SUMMARY:
The purpose of this study was to determine whether TH9507, a stabilized analogue of growth hormone-releasing factor (GRF), would have an effect on insulin sensitivity or control of diabetes in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal or surgically sterilized female subjects, 50 years of age or older;
* Documented diagnosis of type 2 diabetes as defined by the American Diabetes Association;
* Diagnosis of type 2 diabetes for at least 3 months before screening;
* Subjects on stable diabetes treatment regimens (receiving oral hypoglycemics with or without insulin) for at least 2 months before screening;
* Screening and pre-randomization glycosylated hemoglobin (HbA1c) <10.0%, according to central laboratory;
* Body mass index (BMI) between 25 and 38 kg/m2
* Subjects willing to perform specified home blood glucose monitoring and comply with all study protocol requirements;
* Signed informed consent.

Exclusion Criteria:

* Serum creatinine >2 mg/dL;
* Fasting triglycerides >1000 mg/dL;
* Albuminuria >200 mg/24 hours;
* Positive mammography (if female) or prostate-specific antigen (PSA) or prostate examination for cancer (if male);
* Use of oral or parenteral glucocorticoids in the 30 days before screening;
* Use of any experimental or marketed growth hormone, growth hormone secretagogues, insulin-like growth factor-1 (IGF-1), or insulin-like growth factor binding protein-3 (IGFBP-3) during the previous 6 months;
* Subjects with two or more severe hypoglycemia episodes within the past 6 months, or any hospitalization or emergency room visit due to poor glycemic control within the past 6 months. Similarly, during the lead-in period, any subject with more than one severe hypoglycemic episode or any hospitalization or emergency room visit due to poor glycemic control will be excluded from randomization;
* History of or presence of active concomitant conditions or diseases (e.g., myocardial infarction, poorly controlled hypertension, thyroid disease, rheumatoid arthritis, seizure disorder, diabetic neuropathy, diabetic retinopathy [except subjects with only microaneurysms on fundus examination]) that would interfere with the protocol conduct and endpoint measurements;
* Subjects with a major surgical operation during the 30 days before screening;
* Subjects with known hypopituitarism, history of pituitary tumor/surgery, head irradiation, or severe head trauma;
* Current cancer or history of cancer, except non-melanomatous skin cancer;
* Subjects with active infection at any body site or a history of severe infection (requiring oral or parenteral treatment) during the 30 days before screening;
* Subjects with clinically significant abnormalities on screening laboratory evaluation (unless discussed with and approved by the medical monitor);
* Subjects with allergy to synthetic growth hormone products or their excipients;
* Subjects who had previously received growth hormones in any clinical trial;
* Participation in a trial of an experimental drug or device within 90 days before screening.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2002-02; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in relative insulin response

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin (HbA1c)
Change in mean daily serum glucose concentrations
  Home blood glucose will be obtained four times per day (before breakfast, lunch, and dinner, and at bedtime) using a standard blood glucose meter
Changes in the number of dose adjustments per week for insulin and/or oral hypoglycemic agents
Number of subjects with a change in the control of diabetes

REFERENCES:
- [Derived] Clemmons DR, Miller S, Mamputu JC. Safety and metabolic effects of tesamorelin, a growth hormone-releasing factor analogue, in patients with type 2 diabetes: A randomized, placebo-controlled trial. PLoS One. 2017 Jun 15;12(6):e0179538. doi: 10.1371/journal.pone.0179538. eCollection 2017. PMID 28617838